CLINICAL TRIAL: NCT06791798
Title: Effects of Ventilator Hyperinflation Versus Vibrocompression on Lung Compliance in Mechanically Ventilated Patients
Brief Title: Effects of Ventilator Hyperinflation Versus Vibrocompression in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadia Hassan Mohamed Hussien, Physical Therapist, MSc in Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005560
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Mechanically Ventilated Patients; Lung Compliance; Airway Clearance Impairment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study Group (A) (Active Comparator): The patients in the study group (A) will be treated with ventilator hyperinflation in addition to a traditional chest physical therapy program (percussion, postural drainage, and suction) for 4 successive sessions at a rate of one session per day.
  Interventions: Other: Ventilator Hyperinflation; Other: Traditional Chest Physical Therapy Program
- Study Group (B) (Active Comparator): The patients in the study group (B) will be treated with vibrocompression in addition to a traditional chest physical therapy program (percussion, postural drainage, and suction) for 4 successive sessions at a rate of one session per day.
  Interventions: Other: Vibrocompression; Other: Traditional Chest Physical Therapy Program
- Control Group (C) (Active Comparator): The patients in the control group (C) will be treated with a traditional chest physical therapy program (percussion, postural drainage, and suction) for 4 successive sessions at a rate of one session per day.
  Interventions: Other: Traditional Chest Physical Therapy Program

INTERVENTIONS:
Other: Ventilator Hyperinflation — In ventilator hyperinflation volume control mode, the ventilator will be set to eight breaths per minute, and the tidal volume will be increased to deliver hyperinflation breaths that are 15 ml/kg, as will be calculated using the predicted body weight. Tidal volume will be increased in 150-ml increments until a peak airway pressure of 40 cmH2O is achieved. Once this pressure is reached, eight mechanical breaths will be delivered to the patient. After this, the ventilator will be reset to pretreatment variables, and the patient will be rested for 30 s. The sequence will be repeated. The treatment will consist of five sets of eight ventilator hyperinflation breaths.
  Arms: Study Group (A)
Other: Vibrocompression — Vibrocompression will be performed by the physical therapist to produce vibration and will be combined with compression of the patient's chest in the expiratory phase. Every vibrocompression will be interrupted at the end of each expiratory phase to allow free inspiration.
  Arms: Study Group (B)
Other: Traditional Chest Physical Therapy Program — Percussion, Postural Drainage, and Suction

SUMMARY:
The aim of the current study is to compare the effects of ventilator hyperinflation and vibrocompression on lung compliance in mechanically ventilated patients.

DETAILED DESCRIPTION:
Lower respiratory infections remained the world's most deadly communicable disease, ranked as the 4th leading cause of death.

The aim of mechanical ventilation is to reduce the ventilatory work and maintain gas exchange, but it also has deleterious effects on mucociliary transport and coughing ability. These effects provoke the stasis of secretions in the airways and bronchial obstruction, with hypoventilation, atelectasis, and consequent hypoxemia. This set of factors also favors microorganism multiplication and, thus, an increased incidence of ventilator-associated pneumonia (VAP), impaired gas exchange, pulmonary infection and fibrosis, and progressive reduction of lung compliance. To reverse or reduce these deleterious effects, bronchial hygiene techniques are used by physical therapists in several ICUs around the world. Among these techniques, tracheal aspiration, vibrocompression (VB), and hyperinflation with mechanical ventilation are commonly employed.

Lung compliance is inversely proportional to elastance. This elastic resistance is due to the elastic property of lung tissue or parenchyma and the surface elastic force. Any changes occurring to these forces could lead to changes in compliance. Compliance determines 65% of the work of breathing. If the lung has low compliance, it requires more work from breathing muscles to inflate the lungs. In specific pathologies, continuous monitoring of the lung compliance curve is useful to understand the condition's progression and to decide on therapeutic settings needed for ventilator management So, the current study will help to determine the effects of ventilator hyperinflation and vibrocompression on lung compliance and sputum production in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Eighty-one mechanically ventilated patients more than 48 hours up to 7 days
* Their ages range from 35 to 55 years old.
* Medical stability (mean arterial pressure > 60 < 110, systolic blood pressure > 80, diastolic blood pressure > 60, fraction of inspired oxygen < 60, positive end expiratory pressure (PEEP) <10)

Exclusion Criteria:

Patients will be excluded if they have the following conditions or diseases:

* Unstable hemodynamics
* Fraction of inspired oxygen (FiO2) ≥ 0.6
* PEEP ≥ 10 cmH2O
* undrained pneumothorax and hemothorax or subcutaneous emphysema
* Pulmonary pathology (e.g., acute respiratory distress syndrome, exacerbation of chronic obstructive pulmonary disease, and acute pulmonary edema)
* Unstable neurological problems (raised intracranial pressure).
* Lung Cancer
* Recent/unhealed rib fracture
* Any disease obstructs our study.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Static Compliance | Before, after treatment at Day 1 and Day 4
  Static compliance (ml/cmH2O).
Airway Resistance | Before, after treatment at Day 1 and Day 4
  Airway Resistance (cmH2O/l/s).
Sputum Volume in ml | Immediately after treatment at Day 1 and Day 4
  Airway suction will be carried out immediately after treatment or during treatment if indicated and will be measured as sputum volume in ml.
Peak Expiratory Flow and Peak Inspiratory Flow | Before, after treatment at Day 1 and Day 4
  Peak Expiratory Flow (l/min) and Peak Inspiratory Flow (l/min)

SECONDARY OUTCOMES:
Oxygen Saturation (SPO2) | Before, after treatment at Day 1 and Day 4
  Peripheral oxygen saturation (SPO2) in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nadia H Mohamed, MSc, Principal Investigator — Cairo University
Locations (1):
- Kasr AL Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No